CLINICAL TRIAL: NCT02227043
Title: Study Of Adipose Tissue Function and Weight Development Over Time
Brief Title: Study Of Weight Development Over Time
Acronym: SOWOT
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Mikael Ryden, MD, PhD, Professor, Karolinska Institutet
Other Study IDs: SOWOT
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Insulin Resistance; Weight Reduction; Weight Gain
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, adipose tissue, adipocytes
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will study the influence of fat cell size/number and adipose function on weight development over very long time periods (years). By comparing fat biopsies obtained at baseline and after >7 years, the investigators will determine the association between adipose morphology/function and changes in weight or development of cardiometabolic complications (e.g. insulin resistance, type 2 diabetes, dyslipidemia and hypertension).

DETAILED DESCRIPTION:
The investigators will ask all subjects that have previously been examined at the investigators laboratory (from 1992 and forward) in studies of adipose tissue function if they are interested to participate in a new study. The minimal follow up time is 7 years.

Saved blood samples and samples from old fat biopsies will be analyzed together with samples from new examinations.

The investigators plan to examine the subjects in the same way as performed at the baseline examinations. This includes estimation of total body fat using bioimpedance, venous blood samples for determination of insulin, glucose and lipids, subcutaneous fat biopsies with determination of fat cell size/number, lipolysis/lipogenesis as well as analysis of adipokine secretion.

In selected patients, baseline examinations included DEXA-measurement (dual energy x-ray absorptiometry) for determination of body fat distribution as well as hyperinsulinemic euglycemic clamp. In these cases, the same type of examinations will be repeated at their follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Participated in previous examination at our lab at least 7 years ago.
* No blood samples or adipose samples saved from last examination

Exclusion Criteria:

* Decline to participate after invitation.
* Serious illness or mental disorder.
* Warfarin or other new oral anticoagulant that increase risk of bleeding.

Ages: 24 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Observational study All subjects that have been previously investigated at our lab at least 7 years ago
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Weight development over time and correlation to adipose morphology | from 2014 up to 2024, up to 10 years
  Recruitment of these subjects will continue until 2024 with a minimum follow up time of 7 years (84 months). Weight will be assessed with a regular scale and adipose morphology will be determined by measurement of fat cell size and adjustment for body weight.
Weight development and correlation to lipolysis | 2014 to 2024, up to 10 years
  Recruitment of these subjects will continue until 2024 with a minimum follow up time of 7 years. Weight will be assessed with a regular scale. Fat cells will be isolated and assessment of lipolysis will be made with previously published standardized protocols.
Weight development and correlation to lipogenesis | 2014 to 2024, up to 10 years
  Recruitment of these subjects will continue until 2024 with a minimum follow up time of 7 years. Weight will be assessed with a regular scale and lipogenesis will be measured according to previously published standardized protocol after isolated fat cells have been stimulated with insulin.

SECONDARY OUTCOMES:
adipose tissue morphology development and insulin sensitivity | 2014 to 2024, up to 10 years
  Recruitment of these subjects will continue until 2024 with a minimum follow up time of 7 years. Adipose morphology will be determined by measurement of fat cell size and adjustment for body weight. Insulin sensitivity will be assessed by measurement of glucose and insulin and in some cases also hyperinsulinemic euglycemic clamp.
adipose morphology and changes in fat mass | 2014 to 2024, up to 10 years
  Recruitment of these subjects will continue until 2024 with a minimum follow up time of 7 years. Adipose morphology will be determined by measurement of fat cell size and adjustment for body weight. Fat mass will be assessed by impedance measurement and in some cases DEXA according to previously published protocols.
adipose morphology and development of fat mass | 2014 to 2024, up to 10 years
  Recruitment of these subjects will continue until 2024 with a minimum follow up time of 7 years. Fat mass will be assessed by impedance measurement and in some cases DEXA according to previously published protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Ryden, MD, PhD, Principal Investigator — Karolinska Institutet; Peter Arner, MD, PhD, Study Director — Karolinska Institutet; Daniel P Andersson, MD, Study Chair — Karolinska Institutet
Locations (1):
- Lipid laboratory Karolinska University Hospital Huddinge, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Ryden M, Gao H, Arner P. Influence of Aging and Menstrual Status on Subcutaneous Fat Cell Lipolysis. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz245. doi: 10.1210/clinem/dgz245. PMID 31784744
- [Derived] Arner P, Andersson DP, Backdahl J, Dahlman I, Ryden M. Weight Gain and Impaired Glucose Metabolism in Women Are Predicted by Inefficient Subcutaneous Fat Cell Lipolysis. Cell Metab. 2018 Jul 3;28(1):45-54.e3. doi: 10.1016/j.cmet.2018.05.004. Epub 2018 May 31. PMID 29861390